CLINICAL TRIAL: NCT03723382
Title: Stroke in Egyptian Clinical REgisTry
Acronym: SECRET
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Society of Minimally Invasive Neurological Therapeutic Procedures (Network)
Collaborators: Egyptian Stroke Society (Other); Egyptian Society of Neurological Surgeons (Other); Egyptian Radiology Society (Other); Middle East North Africa Stroke and Interventional Neurotherapies Organization (Other)
Responsible Party: Principal Investigator, Prof. Ossama Mansour, Prof of neurology alexandria university, University of Alexandria
Other Study IDs: ESS015000
Record Dates: First submitted 2018-10-07; First posted 2018-10-29 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Stroke, Cardiovascular; Stroke, Acute; Stroke Hemorrhagic; Stroke Spinal Cord; Stroke, Complication
MeSH Terms: conditions — Myocardial Infarction; Stroke; Hemorrhagic Stroke | interventions — Rehabilitation; Secondary Prevention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with stroke with structured management: Patients with the Acute Brain injury, Transient Ischemic Attack, Acute and Chronic Ischemic and Hemorrhagic Stroke, Subarachnoid hemorrhage, and cerebral venous thrombosis from pre-hospitalization, hospitalization (in-patient) and post hospitalization (clinic) data
  Interventions: Other: SECRET structured 5 bundles of standard healthcare services
- Patients with stroke without structured management: Control subject who have stroke and did not managed according to the SECRET 6 level metrics

INTERVENTIONS:
Other: SECRET structured 5 bundles of standard healthcare services — THE 5 BUNDLES OF Stroke SERVICE They the mix of the services for stroke patient which are available at the SS EVT bundle: is the availability of the Endovascular services Telemedicine core bundle : is the ability to guide or guided via tele-medicine for decision making for stoke patients tPA core bundle : the availability of all infrastructure to administer tPA in the first 3 hours of onset (NNT=8) DISMAST bundle : which refer to the availability of Dysphagia detection and management ,Aspirin in hyper acute phase , The Mobilization plans and programs for the patients, anticoagulant and statin prescription for selected patients for secondary prophylaxis programs Process of care bundle : like registering patients and morphology of the disease, screening programs for risk factors , following primary prevention plans all bundles should be judged by the 8M approach
  Other Names: Iv-Thrombolysis; Endovascular treatment; Rehabilitation , mobilization , bulbar care, secondary prevention; Stroke unit calibration; Prehospital care organization
  Groups: Patients with stroke with structured management

SUMMARY:
This is a multi-institutional registry database for the patients with stroke and cerebrovascular diseases. Stroke is the second leading cause of death in the Egypt. Despite extensive research, most of the patients die or suffer from varying degree of post-stroke disabilities due to neurologic deficits.

This registry aims to understand the disease and examine the disease dynamics at the National Level. additionally it aim to introduce an objective method for classifying the registered hospital on a spectrum of 6 level coded with colors (from Black to Green ) according the availability of the predetermined 5 bundles of services presented for patient

DETAILED DESCRIPTION:
A clinical registry is an observational database, usually focusing on a clinical condition, procedure, therapy, or population. A stroke registry can be defined as "an organized system for the collection, storage, retrieval, analysis, and dissemination of information on individual patients who have had a stroke".

An ideal stroke registry is nationwide and enrolls patients from as many participating hospitals as possible in order to increase representativeness and avoid selection bias. For example, the Risk-Stroke register in Sweden, launched in 1994, has covered all hospitals that admit acute stroke patients across the country since 1998 . Appropriate data structure and governance policies are needed to keep a nationwide stroke registry sustainable and operating well. Through the publication and communication of results, a stroke registry should be helpful for improvement of stroke care quality, health policy, and the outcomes of patients.

SECRET registry aim to help in the following

1. National Grading of The Presented Stroke Care Services:

   where A 6 levels grading system was designed according to the capability of each service spot (hospital, center, etc.) to present a range of the 5 stroke service bundles of care. each Service Spot (SS) will have one of the following colors according to the availability of the services.
2. Cost-effectiveness registry Based SOPs SECRET is the first of its type registry to study the parameters for cost/effectiveness analysis for specific steps in the chain of care for stroke patient. The only convincing tool which could be used to approach the politics to be attentive and malleable for changing national plans of healthcare.
3. Aneurysm Registry This Part of the registry is dedicated for the cerebral aneurysm disorders and their type of clinical presentation. The options of treatment and each option effectiveness and cost outcome.

CFD for Best Medical Treatment Registry To investigate the possible application collected from CFD analysis in special situation to guide physician for best medical treatment (BMT) option for a Neurovascular Disorder.

ELIGIBILITY:
Inclusion Criteria:

* All patients with a diagnosis of Acute Brain injury, Transient Ischemic Attack, Acute and Chronic Ischemic and Hemorrhagic Stroke, Subarachnoid hemorrhage, and cerebral venous thrombosis seen in the registered Centers.
* Age > 1 years of age.

Exclusion Criteria:

* Patients who don't have the diagnosis of Acute Brain injury, Transient Ischemic Attack, Acute and Chronic Ischemic and Hemorrhagic Stroke, Subarachnoid hemorrhage, and cerebral venous thrombosis.
* Patients who have Epidural Hematoma, Subdural hematoma.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a final/discharge diagnosis of stroke or transient ischemic attack can be included into the SECRET Registry.
  This includes cases with a principal/primary or secondary diagnosis of:
  Cerebral Infarction Intracerebral Hemorrhage (non-traumatic) Ischemic Stroke Subarachnoid Hemorrhage (non-traumatic) Transient Ischemic Attack (TIA) Cerebral Venous Sinus Thrombosis The investigators will use the available EMR and databases to search for these patients using relevant ICD-9/10 codes. or any other method used internally to archive stroke cases
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2018-05-20 (Actual); Primary Completion 2020-05-19 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
The National Institutes of Health Stroke Scale (NIHSS) reported | 30 days post discharge from hospital
  Severity of ischemic stroke and stroke not otherwise specified patients will be weighted with a score reported for NIH Stroke Scale will be grouped into Mild stroke (>0-6 on NIHSS) moderate (>6 - 10 on NIHSS) severe (>10 - 20 on NIHSS) and Grave (>20 on NIHSS)
Modified Rankin Scale at Discharge | 90 days post discharge from hospital
  Patients grouped by Modified Rankin Scale at discharge
Risk-Adjusted Mortality Ratio for Ischemic-Only and Ischemic and Hemorrhagic models | 30 days post discharge from hospital
  A ratio comparing the actual in-hospital mortality rate to the risk-adjusted expected mortality rate.

SECONDARY OUTCOMES:
Disease burden | 1 year
  Quality-Adjusted Life-Years (QALY) : measure of the life expectancy corrected for loss of quality of that life caused by diseases and disabilities.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University , School of medicine , Neurology Department, Neurovascular Unit, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: once start for 7 years
Access Criteria: registred user to Site Data Non registered User to Stat Data
URL: http://www.strokeregistry.eg

REFERENCES:
- See also: registry website — http://www.strokesregistry.com